CLINICAL TRIAL: NCT04707781
Title: Clinical Database for the Early Recognition of Pulmonary Parenchymal Involvement in Patients With Systemic Diseases Bearing a Risk for Interstitial Lung Disease
Brief Title: Database for Interstitial Lung Disease
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 33-023 ex 20/21
Record Dates: First submitted 2021-01-12; First posted 2021-01-13 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Lung Diseases, Interstitial
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum samples of prospectively included patients will be stored in the Biobank Graz
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- prospective patient cohort: patients who will undergo the prospective ILD Screening algorithm
  Interventions: Diagnostic Test: chest CT
- retrospective patient cohort: patients with diagnosed ILD
  Interventions: Diagnostic Test: chest CT

INTERVENTIONS:
Diagnostic Test: chest CT — assessment of interstitial lung disease using chest CT

SUMMARY:
The purpose of this study is to establish a clinical database for patients bearing at risk for ILD (Interstitial Lung Disease) and to set up a prospective ILD Screening program for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years
* patients with a known systemic disease bearing a risk for ILD
* signed informed consent (for prospective part)

Exclusion Criteria:

* Age < 18 years
* comorbidities severely limiting life-expectancy (e.g. severe cardiovascular conditions, malignant disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (females and males; above 18 yrs) with a known systemic disease bearing a risk for ILD but without diagnosed ILD and patients (females and males; above 18 yrs) with diagnosed ILD.
Sampling Method: Non-Probability Sample
Enrollment: 412 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
DLCO%pred (carbon monoxide diffusing capacity) at time of ILD diagnosis | 5 years
  The investigators aim to assess DLCO% pred at time of ILD diagnosis in patients undergoing a ILD Screening algorithm and compare to the retrospective patient cohort with diagnosed ILD and the DLCO%pred at time of ILD diagnosis

SECONDARY OUTCOMES:
FVC%pred (Forced vital capacity) at time of ILD diagnosis | 5 years
  The investigators aim to assess FVC% pred at time of ILD diagnosis in patients undergoing a ILD Screening algorithm and compare to the retrospective patient cohort with diagnosed ILD and the FVC%pred at time of ILD diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Department of Internal Medicine, Division of Pulmonology, Graz, Austria

IPD SHARING:
Plan to Share IPD: Undecided